CLINICAL TRIAL: NCT00331487
Title: Pioglitazone Versus Rosiglitazone in Subjects With Type 2 Diabetes Mellitus and Dyslipidemia
Brief Title: Study to Compare Pioglitazone and Rosiglitazone in Subjects With Type 2 Diabetes Mellitus and Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H6E-US-GLAI; U1111-1115-9039 (Registry Identifier: WHO)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Pioglitazone; Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone QD (Experimental)
  Interventions: Drug: Pioglitazone
- Rosiglitazone QD (Active Comparator)
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30 mg capsules, orally, once daily and placebo-matching capsules, orally, once daily for up to 12 weeks; increasing to pioglitazone 45 mg, capsules, orally, once daily and placebo-matching capsules, orally, once daily for up to 12 weeks
  Other Names: Actos; AD4833
  Arms: Pioglitazone QD
Drug: Rosiglitazone — Rosiglitazone 4 mg capsules, orally, once daily and placebo-matching capsules, orally, once daily for up to 12 weeks; increasing to rosiglitazone 4 mg, capsules, orally, twice daily for up to 12 weeks
  Arms: Rosiglitazone QD

SUMMARY:
Efficacy comparison of Pioglitazone, once daily (QD), to Rosiglitazone in participants with Type 2 Diabetes

DETAILED DESCRIPTION:
At least two metabolic defects contribute to the development of type 2 diabetes mellitus: relative insulin insufficiency and insulin resistance. The majority of patients with type 2 diabetes mellitus demonstrate some degree of insulin resistance. Even in the absence of hyperglycemia (high blood sugar), insulin resistance is associated with a cluster of metabolic abnormalities that increase the risk for cardiovascular disease, including dyslipidemia (unhealthy blood fat), increased expression of inflammatory markers, activation of pro-coagulants (pro-clotting), hemodynamic changes, and endothelial dysfunction.

The dyslipidemia associated with insulin resistance and type 2 diabetes mellitus is characterized by elevated triglyceride levels and decreased high-density lipoprotein (good) cholesterol levels. Although low-density lipoprotein (bad) cholesterol levels may not be significantly elevated in patients with type 2 diabetes mellitus, an increase in the proportion of small, dense low-density lipoprotein cholesterol particles of increased atherogenicity (increased formation of lipid deposits in the arteries) is observed. When compared with individuals without type 2 diabetes mellitus, the risk of cardiovascular disease is 2- to 4-fold greater in patients with type 2 diabetes mellitus, and the dyslipidemia of diabetes is an important contributor to the increased risk in this population.

By targeting the insulin resistance underlying type 2 diabetes mellitus, the thiazolidinedione class of oral antihyperglycemic medications possesses both a glucose-lowering effect and the potential to alter lipid/lipoprotein metabolism. Two thiazolidinediones are currently available for the treatment of type 2 diabetes mellitus: pioglitazone hydrochloride (ACTOS, Takeda Pharmaceuticals North America, Inc, Lincolnshire, IL) and rosiglitazone maleate (Avandia, GlaxoSmithKline, Research Triangle Park, NC).

The purpose of this study is to evaluate the triglyceride-lowering effects of pioglitazone to rosiglitazone in patients with type 2 diabetes mellitus and dyslipidemia who are not receiving any other glucose- or lipid-lowering therapies at the same time as the study medications.

Individuals who participate in this study will provide written informed consent and will be required to commit to a screening visit and approximately 7 additional visits at the study center. Study participation is anticipated to be about 39 weeks (or approximately 8 months). Multiple procedures will occur at each visit which may include fasting, blood collection, physical examinations and electrocardiograms. Participants will be required to follow a diabetic diet, self-monitor their blood glucose and maintain a study diary for the duration of the study.

ELIGIBILITY:
Inclusion Criteria

* Type 2 diabetes mellitus according to the World Health Organization criteria and have diabetes-associated dyslipidemia (fasting triglycerides level between greater than or equal to 150 mg per dL and less than or equal to 600 mg per dL, and a fasting direct low-density lipoprotein cholesterol less than or equal to 130 mg per dL).
* Fasting serum C-peptide greater than or equal to1 ng per
* Glycosylated hemoglobin greater than or equal to 7% and less than or equal to 11% if naive to oral antihyperglycemic medications, or greater than or equal to 9.5% if previously treated with oral antihyperglycemic monotherapy

Exclusion Criteria

* Investigator site personnel and their immediate families. Immediate family defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Treatment with a drug within 30 days of Visit 1 that had not received regulatory approval.
* Treatment within 60 days of Visit 1 with any of the following:

  * insulin
  * systemic glucocorticoid therapy (excluding topical and inhaled preparations)
  * combination glycemic therapy (two or more oral anti-diabetes medications)
  * any lipid-lowering agent (including nicotinic acid, fibrates, bile acid resin binders, statins, d thyroxine or neomycin)
  * any weight loss agent (prescription or over the counter)
* Pregnant, breast feeding, or intending to become pregnant during the study.
* Serum creatinine greater than or equal to 176.8 μmol per L or greater than or equal to 2 plus per dipstick.
* Proteinuria at Visit 1.
* Alanine transaminase or aspartate transaminase greater than or equal to 1.5 times the upper limit of normal at Visit 1 or had significant clinical signs or symptoms of liver disease.
* History of signs or symptoms of liver disease, such as jaundice or alanine transaminase greater than or equal to 1.5 times the upper limit of normal, while treated with any thiazolidinedione
* Hemoglobin less than 10.5 g per dL for females and less than11.5 g per dL for males at Visit 1.
* Clinically or biochemically based on thyroid stimulating hormone at Visit 1 hypothyroid or hyperthyroid.
* History of myocardial infarction, acute cardiovascular event, or heart surgery within 6 months of Visit 1.
* Functional New York Heart Association Cardiac Class III or IV disease.
* Receiving renal dialysis or has had received a renal transplant.
* Undergoing therapy for a malignancy other than basal cell or squamous cell skin cancer.
* Clinical signs or symptoms of drug or alcohol abuse.
* History of HIV infection.
* Allergy to any glitazone drug.
* Medical history or the presence of any clinically significant or unstable medical condition that made the patient unlikely to complete the study.
* Any condition or situations that precluded adherence and completion of the protocol or a precluding ability to voluntarily give informed consent.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2000-09; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Change in fasting triglyceride level | Final Visit

SECONDARY OUTCOMES:
Change in fasting low-density lipoprotein cholesterol. | Final Visit
Change in fasting high-density lipoprotein cholesterol. | Final Visit
Change in fasting total cholesterol. | Final Visit
Change in fasting free fatty acids. | Final Visit
Change in plasminogen activator inhibitor 1 | Final Visit
Change in high-sensitivity C-reactive protein | Final Visit
Change in fasting C-peptide. | Final Visit
Homeostasis model assessment-insulin resistance mode. | Final Visit
Change in fasting insulin. | Final Visit
Homeostasis model assessment-beta cell function. | Final Visit
Change in glycosylated hemoglobin. | Final Visit
Change in fasting plasma glucose. | Final Visit
Low-density lipoprotein particle concentration. | Final Visit
Low-density lipoprotein particle size. | Final Visit
High-density lipoprotein particle size. | Final Visit
Very low-density lipoprotein particle size. | Final Visit
Apolipoprotein A-I. | Final Visit
Apolipoprotein B | Final Visit
Lipoprotein a | Final Visit
Apolipoprotein C-III. | Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Perez, MD, Study Director — Takeda
Locations (66):
- United States (66):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Tucson, Arizona
  - Concord, California
  - Fremont, California
  - Los Angeles, California
  - Palos Verdes Estates, California
  - San Diego, California
  - Santa Barbara, California
  - Santa Rosa, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Avon, Connecticut
  - Hamden, Connecticut
  - Longwood, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Fayetteville, Georgia
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - South Bend, Indiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Frederick, Maryland
  - Salisbury, Massachusetts
  - South Yarmouth, Massachusetts
  - Waltham, Massachusetts
  - Minneapolis, Minnesota
  - Chesterfield, Missouri
  - Omaha, Nebraska
  - East Setauket, New York
  - Endwell, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Morehead City, North Carolina
  - Wilmington, North Carolina
  - Columbus, Ohio
  - Franklin, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Salem, Oregon
  - Philadelphia, Pennsylvania
  - Pottstown, Pennsylvania
  - Providence, Rhode Island
  - Mt. Pleasant, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Beaumont, Texas
  - Conroe, Texas
  - Dallas, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Mechanicsville, Virginia
  - Newport News, Virginia
  - Virginia Beach, Virginia
  - Federal Way, Washington
  - Wenatchee, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Goldberg RB, Kendall DM, Deeg MA, Buse JB, Zagar AJ, Pinaire JA, Tan MH, Khan MA, Perez AT, Jacober SJ; GLAI Study Investigators. A comparison of lipid and glycemic effects of pioglitazone and rosiglitazone in patients with type 2 diabetes and dyslipidemia. Diabetes Care. 2005 Jul;28(7):1547-54. doi: 10.2337/diacare.28.7.1547. PMID 15983299
- [Result] Tilden DP, Mariz S, O'Bryan-Tear G, Bottomley J, Diamantopoulos A. A lifetime modelled economic evaluation comparing pioglitazone and rosiglitazone for the treatment of type 2 diabetes mellitus in the UK. Pharmacoeconomics. 2007;25(1):39-54. doi: 10.2165/00019053-200725010-00005. PMID 17192117
- [Result] Deeg MA, Buse JB, Goldberg RB, Kendall DM, Zagar AJ, Jacober SJ, Khan MA, Perez AT, Tan MH; GLAI Study Investigators. Pioglitazone and rosiglitazone have different effects on serum lipoprotein particle concentrations and sizes in patients with type 2 diabetes and dyslipidemia. Diabetes Care. 2007 Oct;30(10):2458-64. doi: 10.2337/dc06-1903. Epub 2007 Jun 26. PMID 17595355
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI